CLINICAL TRIAL: NCT00327821
Title: A Randomised Control Trial of Commercial Weight Loss Programme in a Community Based Sample of Obese Adults.
Brief Title: The Effectiveness of Commercial Weight Loss Programmes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: British Broadcasting Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 107189 BBC
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2003-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

INTERVENTIONS:
Behavioral: calorie controlled diet

SUMMARY:
The objective is to compare the effectiveness of 4 different commercial weight-loss diets available to adults in the UK.

This is achieved with a 6 month multi-centre randomised unblinded controlled trial of

* Dr Atkins' New Diet Revolution,
* The slimFast Plan,
* The weight Watchers Pure Points Programme,
* Rosemary Conley's "Eat Yourself Slim" Diet & Fitness Plan.
* No diet (control)

Subjects are a community based sample of 300 (60 per group) otherwise healthy overweight and obese adults.

Main outcome measures are weight and body fat change over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 27 and < 40 kg/m2.

Exclusion Criteria:

* History of coronary heart disease
* Type 1 or Type 2 diabetes
* Renal, liver or respiratory failure
* Gout
* Taking lipid lowering or anti-hypertensive drugs
* History of obesity with known cause (i.e. Cushings disease, hypothyroidism)
* Previous gastric or weight loss surgery
* Taking any weight loss drug (including Orlistat or Sibutramine)
* Clinical depression
* Eating disorders
* Drug or alcohol abuse
* Any malabsorptive state (including lactose intolerance)
* Being treated for a malignancy
* Being pregnant
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-07; Study Completion 2003-03

PRIMARY OUTCOMES:
Weight loss
Fat loss

CONTACTS AND LOCATIONS:
Overall Officials: D J Millward, PhD, Principal Investigator — University of Surrey; H A Truby, PhD SRD, Study Director — University of Surrey
Locations (1):
- University of Surrey, Guildford, surrey, United Kingdom

REFERENCES:
- [Result] Truby H, Baic S, deLooy A, Fox KR, Livingstone MB, Logan CM, Macdonald IA, Morgan LM, Taylor MA, Millward DJ. Randomised controlled trial of four commercial weight loss programmes in the UK: initial findings from the BBC "diet trials". BMJ. 2006 Jun 3;332(7553):1309-14. doi: 10.1136/bmj.38833.411204.80. Epub 2006 May 23. PMID 16720619
- [Derived] Truby H, Hiscutt R, Herriot AM, Stanley M, Delooy A, Fox KR, Baic S, Robson PJ, Macdonald I, Taylor MA, Ware R, Logan C, Livingstone M. Commercial weight loss diets meet nutrient requirements in free living adults over 8 weeks: a randomised controlled weight loss trial. Nutr J. 2008 Sep 2;7:25. doi: 10.1186/1475-2891-7-25. PMID 18764946